CLINICAL TRIAL: NCT04670458
Title: Derivation of An In-Hospital Cardiac Arrest Prediction Model for Patients in Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: IHCA-EWS-QLH
Record Dates: First submitted 2020-11-26; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: In-Hospital Cardiac Arrest
Keywords: Critically ill patients; In-Hospital Cardiac Arrest; Early recognition; Early warning score

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CA group: Patients with In-Hospital Cardiac Arrest
  Interventions: Other: no intervention
- CONTROL group: Patients without In-Hospital Cardiac Arrest
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Current studies have shown that hospitalized ICU patients have a high risk of IHCA, with an incidence of about 0.6-7.8%. Early prediction of the occurrence of IHCA in severe patients can provide early intervention, prevent the deterioration of the disease, and reduce the incidence of IHCA. Therefore, researchers wanted to verify the efficacy of MEWS, NEWS, and CART scores in predicting IHCA in ICU inpatients, and to establish an early-warning scoring model that could effectively predict the risk of IHCA occurrence in ICU inpatients during hospitalization.

ELIGIBILITY:
CA group

Inclusion Criteria:

* Occurrence of IHCA
* Hospital stay ≥48h.

Exclusion Criteria:

* <14 years
* Do Not Resuscitat
* Patients hospitalized due to out-of-hospital cardiac arrest
* Cardiac arrest occurs during the operation
* The patients with implanted cardiac pacemaker suffered cardiac arrest due to instrument malfunction.

CONTROL group

Inclusion Criteria:

* Without IHCA
* Hospital stay ≥48h

Exclusion Criteria:

* <14 years
* Leave hospital without medical advice

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in the intensive care unit (ICU, CCU, RICU, EICU, NCU and DICU) of Qilu Hospital of Shandong University from January 1, 2017 to October 31, 2019 were selected.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
In-Hospital Cardiac Arrest | Day 2
  Cardiac arrest occurs during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China